CLINICAL TRIAL: NCT04447404
Title: A Randomized, Double-Blind, Placebo Controlled Study to Evaluate Safety and Efficacy of DUR-928 in Subjects Infected With SARS-CoV-2 With Acute Lung, Liver or Kidney Injury
Brief Title: DUR-928 in Subjects With SARS-CoV-2 With Acute Lung, Liver or Kidney Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Durect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C928-020
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Intervention Model Description: 3:1 randomization DUR-928:placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DUR-928 (Experimental)
  Interventions: Drug: DUR-928
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DUR-928 — IV infusion
  Arms: DUR-928
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
Evaluate safety and efficacy of DUR-928 in treatment of acute organ failure in subjects infected with SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with moderate, severe, or early critical COVID-19 illness diagnosed by RT- PCR
* Acute liver injury (including acute on chronic liver disease) or acute kidney injury or moderate COVID-19 pneumonia

Exclusion Criteria:

* Critical COVID-19 illness (MAP < 60 mm Hg, on mechanical ventilator for ≥ 5 days)
* On maintenance hemodialysis or peritoneal dialysis
* Child Pugh C cirrhosis
* Hepatorenal syndrome
* Ascites and/or hepatic encephalopathy
* History of end stage renal disease or CKD with eGFR < 15 mL/min/1.73m2
* Women who are pregnant or breast feeding
* Receipt of other concomitant experimental therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gordon, MD, Study Director — CTI Clinical Trial and Consulting Services
Locations (1):
- Site 03, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DUR-928 | Placebo
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early due to lack of enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | DUR-928 | Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (16.26) |  | 66.5 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of Alive and Free of Organ Failure at Day 28
Description: Free of mechanical ventilation, free of renal replacement therapy and free of acute liver failure
Time Frame: Day 28
Population: Study was terminated early with only 2 subjects enrolled, both assigned to active treatment. Both subject deaths were assessed as Not Related to study treatment occurring on Day 19 and Day 20 (15 and 16 days after last dose, respectively).
Measure: Count of Participants; unit: Participants
Arm/Group | DUR-928 | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

2. Secondary Outcome: Alive at Days 28 and 60
Time Frame: Day 28 and Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DUR-928 | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

3. Secondary Outcome: Alive, Out of ICU, at Day 28
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DUR-928 | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

4. Secondary Outcome: Alive, Out of Hospital, at Days 28 and 60
Time Frame: Day 28 and Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DUR-928 | Placebo
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Description: Due to early study termination, no subjects were enrolled in the placebo treatment group.
Arm/Group | DUR-928 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUR-928 (N=2) | Placebo (N=0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 — ACUTE HYPOXIC RESPIRATORY FAILURE 2/2 COVID PNA 2/2 TERMINAL EXTUBATION
Brain Injury (Nervous system disorders) | 1 (1) | 0 — ANOXIC BRAIN INJURY SECONDARY TO CEREBRAL EDEMA AND SAH
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUR-928 (N=2) | Placebo (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0
Bradycardia (Cardiac disorders) | 1 (1) | 0
Pyrexia (General disorders) | 2 (3) | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (1) | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 0
Hypotension (Vascular disorders) | 2 (2) | 0

LIMITATIONS AND CAVEATS:
Early study termination led to small number (n=2) of subjects and in one treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that if sponsor has not submitted a multi-site publication within 18 months of study completion, the PI can submit the sponsor results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The PI will remove confidential information from results communications prior to publication upon request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04447404/Prot_SAP_001.pdf